CLINICAL TRIAL: NCT01912456
Title: A Double-blind, Randomized, Placebo-controlled, Cross-over Study to Evaluate the Clinical Efficacy and Safety of Subcutaneous Administration of Human Plasma-derived C1-esterase Inhibitor in the Prophylactic Treatment of Hereditary Angioedema
Brief Title: A Study to Evaluate the Clinical Efficacy and Safety of Subcutaneously Administered C1-esterase Inhibitor in the Prevention of Hereditary Angioedema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CSL830_3001; 2013-000916-10 (EudraCT Number)
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Results first posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Hereditary Angioedema Types I and II
Keywords: Hereditary Angioedema
MeSH Terms: conditions — Hereditary Angioedema Types I and II; Angioedemas, Hereditary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Higher-volume placebo, then low-volume C1-esterase inhibitor (Experimental): A higher-volume dose of placebo will be administered subcutaneously twice a week for up to 16 weeks, then a low-volume dose of C1-esterase inhibitor will be administered subcutaneously twice a week for up to 16 weeks.
  Interventions: Biological: Low-volume C1-esterase inhibitor; Biological: Higher-volume placebo
- Low-volume C1-esterase inhibitor, then higher-volume placebo (Experimental): A low-volume dose of C1-esterase inhibitor will be administered subcutaneously twice a week for up to 16 weeks, then a higher-volume dose of placebo will be administered subcutaneously twice a week for up to 16 weeks.
  Interventions: Biological: Low-volume C1-esterase inhibitor; Biological: Higher-volume placebo
- Low-volume placebo, then higher-volume C1-esterase inhibitor (Experimental): A low-volume dose of placebo will be administered subcutaneously twice a week for up to 16 weeks then a higher-volume dose of C1-esterase inhibitor will be administered subcutaneously twice a week for up to 16 weeks.
  Interventions: Biological: Higher-volume C1-esterase inhibitor; Biological: Low-volume placebo
- Higher-volume C1-esterase inhibitor, then low-volume placebo (Experimental): A higher-volume dose of C1-esterase inhibitor will be administered subcutaneously twice a week for up to 16 weeks, then a low-volume dose of placebo will be administered subcutaneously twice a week for up to 16 weeks.
  Interventions: Biological: Higher-volume C1-esterase inhibitor; Biological: Low-volume placebo

INTERVENTIONS:
Biological: Low-volume C1-esterase inhibitor
  Arms: Higher-volume placebo, then low-volume C1-esterase inhibitor; Low-volume C1-esterase inhibitor, then higher-volume placebo
Biological: Higher-volume C1-esterase inhibitor
  Arms: Higher-volume C1-esterase inhibitor, then low-volume placebo; Low-volume placebo, then higher-volume C1-esterase inhibitor
Biological: Low-volume placebo
  Arms: Higher-volume C1-esterase inhibitor, then low-volume placebo; Low-volume placebo, then higher-volume C1-esterase inhibitor
Biological: Higher-volume placebo
  Arms: Higher-volume placebo, then low-volume C1-esterase inhibitor; Low-volume C1-esterase inhibitor, then higher-volume placebo

SUMMARY:
The aim of this study is to assess the efficacy of C1-esterase inhibitor in preventing hereditary angioedema attacks when it is administered under the skin of subjects with hereditary angioedema. The safety of C1-esterase inhibitor will also be assessed. Each subject will enter a run-in period of up to 8-weeks. Subjects who complete the run-in period and who are eligible will then enter the treatment phase which comprises two sequential treatment periods. In the treatment phase, subjects will be randomized to one of four arms consisting of treatment with low- or higher-volume C1-esterase inhibitor in one treatment period and treatment with low- or higher-volume placebo in the other treatment period. The study will measure the number of hereditary angioedema attacks that subjects experience while receiving each treatment.

ELIGIBILITY:
Inclusion Criteria:

Run-In Period Inclusion Criteria:

* Males or females aged 12 years or older.
* A clinical diagnosis of hereditary angioedema type I or II.
* Hereditary angioedema attacks over a consecutive 2-month period that required acute treatment, medical attention, or caused significant functional impairment.
* For subjects who have used oral therapy for prophylaxis against HAE attacks within 3 months of Screening: use of a stable regimen within 3 months of Screening, with no plans to change.

Eligibility Criteria for Entering Treatment Period 1:

* Laboratory confirmation of type I or type II hereditary angioedema, including C1-esterase inhibitor functional activity less than 50% AND C4 antigen level below the laboratory reference range.
* No clinically significant abnormalities as assessed using laboratory parameters.
* During participation in the run-in period, subjects must have experienced hereditary angioedema attacks that required acute treatment, required medical attention, or caused significant functional impairment.

Exclusion Criteria:

Run-In Period Exclusion Criteria:

* History of clinical significant arterial or venous thrombosis, or current history of a clinically significant prothrombotic risk.
* Incurable malignancies at screening.
* Any clinical condition that will interfere with the evaluation of C1-esterase inhibitor therapy.
* Clinically significant history of poor response to C1-esterase therapy for the management of hereditary angioedema.
* Receiving therapy prohibited by the protocol, including medications for hereditary angioedema prophylaxis.
* Female subjects who started taking or changed dose of any hormonal contraceptive regimen or hormone replacement therapy (i.e., estrogen/progesterone-containing products) within 3 months prior to the screening visit.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Program Director, Study Director — CSL Behring
Locations (38):
- United States (19):
  - Study Site, Birmingham, Alabama
  - Study Site, Scottsdale, Arizona
  - Study Site, Bell Gardens, California
  - Study Site, La Jolla, California
  - Study Site, Orange, California
  - Study Site, Walnut Creek, California
  - Study Site, Colorado Springs, Colorado
  - Study Site, Chevy Chase, Maryland
  - Study Site, Boston, Massachusetts
  - Study Site, Cincinnati, Ohio
  - Study Site, Columbus, Ohio
  - Study Site, Toledo, Ohio
  - Study Site, Tulsa, Oklahoma
  - Study Site, Lake Oswego, Oregon
  - Study Site, Hershey, Pennsylvania
  - Study Site, Dallas, Texas
  - Study Site, Richmond, Virginia
  - Study Site, Virginia Beach, Virginia
  - Study Site, Spokane, Washington
- Study Site, Campbelltown, New South Wales, Australia
- Canada (4):
  - Study Site, Hamilton, Ontario
  - Study Site, Ottawa, Ontario
  - Study Site, Toronto, Ontario
  - Study Site, Québec
- Czechia (2):
  - Study Site, Hradec Králové
  - Study Site, Pilsen
- Study Site, Budapest, Hungary
- Israel (2):
  - Study Site, Tel Aviv
  - Study Site, Tel Litwinsky
- Italy (2):
  - Study Site, Catania
  - Study Site, Palermo
- Romania (2):
  - Study Site, Cluj-Napoca
  - Study Site, Mures
- Spain (3):
  - Study Site, Barcelona
  - Study Site, Madrid
  - Study Site, Valencia
- United Kingdom (2):
  - Study Site, Brighton
  - Study Site, London

REFERENCES:
- [Result] Longhurst H, Cicardi M, Craig T, Bork K, Grattan C, Baker J, Li HH, Reshef A, Bonner J, Bernstein JA, Anderson J, Lumry WR, Farkas H, Katelaris CH, Sussman GL, Jacobs J, Riedl M, Manning ME, Hebert J, Keith PK, Kivity S, Neri S, Levy DS, Baeza ML, Nathan R, Schwartz LB, Caballero T, Yang W, Crisan I, Hernandez MD, Hussain I, Tarzi M, Ritchie B, Kralickova P, Guilarte M, Rehman SM, Banerji A, Gower RG, Bensen-Kennedy D, Edelman J, Feuersenger H, Lawo JP, Machnig T, Pawaskar D, Pragst I, Zuraw BL; COMPACT Investigators. Prevention of Hereditary Angioedema Attacks with a Subcutaneous C1 Inhibitor. N Engl J Med. 2017 Mar 23;376(12):1131-1140. doi: 10.1056/NEJMoa1613627. PMID 28328347
- [Derived] Beard N, Frese M, Smertina E, Mere P, Katelaris C, Mills K. Interventions for the long-term prevention of hereditary angioedema attacks. Cochrane Database Syst Rev. 2022 Nov 3;11(11):CD013403. doi: 10.1002/14651858.CD013403.pub2. PMID 36326435
- [Derived] Li HH, Zuraw B, Longhurst HJ, Cicardi M, Bork K, Baker J, Lumry W, Bernstein J, Manning M, Levy D, Riedl MA, Feuersenger H, Prusty S, Pragst I, Machnig T, Craig T; COMPACT Investigators. Subcutaneous C1 inhibitor for prevention of attacks of hereditary angioedema: additional outcomes and subgroup analysis of a placebo-controlled randomized study. Allergy Asthma Clin Immunol. 2019 Aug 28;15:49. doi: 10.1186/s13223-019-0362-1. eCollection 2019. PMID 31485239

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo High/CSL830 (40): High-volume dose of placebo administered subcutaneously twice a week for up to 16 weeks, then a low-volume dose of C1-esterase inhibitor (CSL830, 40 IU/kg) administered subcutaneously twice a week for up to 16 weeks.
- CSL830 (40)/Placebo High: A low-volume dose of C1-esterase inhibitor (CSL830, 40 IU/kg) administered subcutaneously twice a week for up to 16 weeks, then a high-volume dose of placebo administered subcutaneously twice a week for up to 16 weeks.
- Placebo Low/CSL830 (60): A low-volume dose of placebo administered subcutaneously twice a week for up to 16 weeks then a high-volume dose of C1-esterase inhibitor (CSL830, 60 IU/kg) administered subcutaneously twice a week for up to 16 weeks.
- CSL830 (60)/Placebo Low: A high-volume dose of C1-esterase inhibitor (CSL830, 60 IU/kg) administered subcutaneously twice a week for up to 16 weeks, then a low-volume dose of placebo administered subcutaneously twice a week for up to 16 weeks.
Period: Period 1
Arm/Group | Placebo High/CSL830 (40) | CSL830 (40)/Placebo High | Placebo Low/CSL830 (60) | CSL830 (60)/Placebo Low
Started | 22 | 23 | 23 | 22
Completed | 20 | 22 | 21 | 19
Not Completed | 2 | 1 | 2 | 3
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — non-compliance | 1 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1
Period: Period 2
Arm/Group | Placebo High/CSL830 (40) | CSL830 (40)/Placebo High | Placebo Low/CSL830 (60) | CSL830 (60)/Placebo Low
Started | 20 | 22 | 21 | 19
Completed | 20 | 20 | 21 | 18
Not Completed | 0 | 2 | 0 | 1
Not completed — Lack of Efficacy | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CSL830 (40)/Placebo High | CSL830 (60)/Placebo Low | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 4 | 7
  Between 18 and 65 years | 38 | 38 | 76
  >=65 years | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (14.41) | 36.8 (14.921) | 39.6 (14.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 32 | 60
  Male | 17 | 13 | 30
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 5 | 8
  Romania | 1 | 0 | 1
  Hungary | 2 | 2 | 4
  United States | 28 | 26 | 54
  Czechia | 1 | 0 | 1
  United Kingdom | 2 | 1 | 3
  Italy | 2 | 3 | 5
  Israel | 3 | 6 | 9
  Australia | 0 | 1 | 1
  Spain | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: The Time-normalized Number of Hereditary Angioedema Attacks
Description: The time normalized number of HAE attacks as reported by the investigator per subject was calculated as: The total number of HAE attacks per subject and per treatment period / length of stay of subject in treatment period (days), Where length of stay of subject in treatment period was calculated as: Date of last day of subject in treatment period - date of first day of Week 3 of subject in treatment period + 1.
Time Frame: During the treatment phase, up to 28 weeks.
Population: Intention-to-treat (ITT) population consisted of all subjects who provided informed consent / assent and were randomized, regardless of whether they received investigational product.
Measure: Least Squares Mean (Standard Error); unit: attacks/day
Groups:
- CSL830 (40): Low-volume dose of C1-esterase inhibitor (CSL830, 40 IU/kg) administered subcutaneously twice a week for up to 16 weeks.
- CSL830 (60): High-volume dose of C1-esterase inhibitor (CSL830, 60 IU/kg) administered subcutaneously twice a week for up to 16 weeks.
- Placebo High: High-volume dose of placebo administered subcutaneously twice a week for up to 16 weeks
- Placebo Low: Low-volume dose of placebo administered subcutaneously twice a week for up to 16 weeks
Arm/Group | CSL830 (40) | CSL830 (60) | Placebo High | Placebo Low
Number analyzed (Participants) | 43 | 43 | 44 | 42
attacks/day | 0.04 (0.011) | 0.02 (0.009) | 0.12 (0.011) | 0.13 (0.009)
Statistical Analysis 1: Comparison: CSL830 (60) vs Placebo Low; Test type: Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: CSL830 (40) vs Placebo High; Test type: Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 3: Comparison: CSL830 (40) vs CSL830 (60); Test type: Other; p = 0.114, Mixed Models Analysis

2. Secondary Outcome: Percentage of Subjects With a ≥ 50% Reduction in the Number of Hereditary Angioedema Attacks by CSL830 Treatment
Description: The percentage reduction (%) in the time normalized number of HAE attacks was calculated as: 100 x [1 - (the time normalized number of HAE attacks when treated with CSL830) / (the time normalized number of HAE attacks when treated with placebo)]. A subject is classed as a responder if the percentage reduction is >= 50%.
Time Frame: During the treatment phase, up to 28 weeks.
Population: ITT. Subjects whose time-normalized number of attacks could not be calculated in one or both CSL830 treatment periods were excluded from the analysis. Percentages are based on the number of subjects included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CSL830 (40) | CSL830 (60)
Number analyzed (Participants) | 42 | 40
percentage of participants | 76.2 [61.5 to 86.5] | 90.0 [76.9 to 96.0]
Statistical Analysis 1: Comparison: CSL830 (40) vs CSL830 (60); Test type: Other; difference in percentages of responder = 13.8, 95% CI 2-sided [-2.8 to 29.7]

3. Secondary Outcome: Time-Normalized Number of Uses of Rescue Medication
Description: The time-normalized number of uses of rescue medication during treatment with C1-esterase inhibitor or placebo
Time Frame: During the treatment phase, up to 28 weeks.
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: rescue medication uses/day
Arm/Group | CSL830 (40) | CSL830 (60) | Placebo High | Placebo Low
Number analyzed (Participants) | 43 | 43 | 44 | 42
rescue medication uses/day | 0.04 (0.042) | 0.01 (0.011) | 0.18 (0.04) | 0.13 (0.011)
Statistical Analysis 1: Comparison: CSL830 (60) vs Placebo Low; Test type: Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: CSL830 (40) vs Placebo High; Test type: Other; p = 0.018, Mixed Models Analysis
Statistical Analysis 3: Comparison: CSL830 (40) vs CSL830 (60); Test type: Other; p = 0.31, Mixed Models Analysis

4. Secondary Outcome: Percentage of Subjects With Adverse Events (AEs) Within 24 Hours of C1-esterase Inhibitor or Placebo Administration
Time Frame: Within 24 hours of C1-esterase inhibitor or placebo administration.
Population: The Safety Population (SP) consisted of all subjects who provided informed consent / assent, were randomized, and received at least 1 dose (or partial dose) of investigational product.
Measure: Number; unit: percentage of participants
Arm/Group | CSL830 (40) | CSL830 (60) | Placebo High | Placebo Low
Number analyzed (Participants) | 43 | 43 | 44 | 42
percentage of participants | 58.1 | 60.5 | 45.5 | 54.8

5. Secondary Outcome: Percentage of Subjects With AEs or Other Specified Safety Events.
Description: The percentage of subjects experiencing the following during treatment with CSL830 and placebo: unsolicited AEs, serious AEs, suspected adverse drug reactions, increased risk scores for deep vein thrombosis and pulmonary embolism, thromboembolic events, inhibitory anti C1 INH antibodies, or clinically significant abnormalities in laboratory assessments.
Time Frame: During the treatment phase, up to 32 weeks.
Population: SP
Measure: Number; unit: percentage of participants
Arm/Group | CSL830 (40) | CSL830 (60) | Placebo High | Placebo Low
Number analyzed (Participants) | 43 | 43 | 44 | 42
percentage of participants | 67.4 | 69.8 | 61.4 | 71.4

6. Secondary Outcome: Percentage of Subjects Experiencing Solicited AEs (Injection Site Reactions)
Description: The percentage of subjects experiencing solicited local AEs (discomfort [eg, pain, burning], swelling, bruising, or itching at the investigational product injection site) during treatment with CSL830 and placebo.
Time Frame: During the treatment phase, up to 32 weeks.
Population: SP
Measure: Number; unit: percentage of participants
Arm/Group | CSL830 (40) | CSL830 (60) | Placebo High | Placebo Low
Number analyzed (Participants) | 43 | 43 | 44 | 42
percentage of participants | 27.9 | 34.9 | 22.7 | 26.2

7. Secondary Outcome: Injections Resulting in Solicited AEs (Injection Site Reactions)
Description: The rate/injection of injections of C1-esterase inhibitor or placebo that were followed by solicited local AEs (discomfort [eg, pain, burning], swelling, bruising, or itching at the investigational product injection site) during treatment with CSL830 and placebo. Rate/Injection = Number of events/number of injections.
Time Frame: During the treatment phase, up to 32 weeks.
Population: SP
Measure: Number; unit: injection site reactions/injection
Units Other Than Participants: number of injections within treatment
Arm/Group | CSL830 (40) | CSL830 (60) | Placebo High | Placebo Low
Number analyzed (Participants) | 43 | 43 | 44 | 42
Number analyzed (number of injections within treatment) | 1307 | 1320 | 1290 | 1164
injection site reactions/injection | 0.21 | 0.08 | 0.12 | 0.05

ADVERSE EVENTS:
Time Frame: During the treatment phase, up to 32 weeks.
Description: The Safety Population consisted of all subjects who provided informed consent / assent, were randomized, and received at least 1 dose (or partial dose) of investigational product
Arm/Group | CSL830 (40) | CSL830 (60) | Placebo High | Placebo Low
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43 | 0/44 | 0/42
Serious Adverse Events (participants affected / at risk) | 1/43 | 0/43 | 1/44 | 1/42
Other Adverse Events (participants affected / at risk) | 10/43 | 17/43 | 12/44 | 12/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSL830 (40) (N=43) | CSL830 (60) (N=43) | Placebo High (N=44) | Placebo Low (N=42)
Hereditary angioedema (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSL830 (40) (N=43) | CSL830 (60) (N=43) | Placebo High (N=44) | Placebo Low (N=42)
Dizziness (Nervous system disorders) | 4 (5) | 0 (0) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 7 (86) | 9 (20) | 6 (36) | 7 (28)
Injection site pain (General disorders) | 7 (90) | 7 (19) | 5 (34) | 4 (9)
Injection site bruising (General disorders) | 2 (5) | 4 (5) | 2 (2) | 3 (5)
Injection site swelling (General disorders) | 1 (1) | 4 (39) | 2 (6) | 2 (18)
Injection site induration (General disorders) | 3 (8) | 4 (6) | 1 (2) | 1 (2)
Fatigue (General disorders) | 1 (1) | 1 (1) | 3 (3) | 3 (3)
Injection site edema (General disorders) | 5 (60) | 0 (0) | 2 (62) | 1 (1)
Injection site haemorrhage (General disorders) | 3 (8) | 1 (1) | 4 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (4) | 2 (4)
Nasopharyngitis (Infections and infestations) | 1 (1) | 8 (9) | 3 (3) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.